CLINICAL TRIAL: NCT07380477
Title: CSF Lactate and Ventriculostomy Associated Infections in Patients With Acute Brain Injury - a Prospective, Observational Cohort Study.
Brief Title: VentricuLostomy AssoCiaTed InfeCtions (LACTIC): Focus on CSF Lactate and Sampling Site
Acronym: LACTIC
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pernille Rosenfeldt, MD, PhD-student, Rigshospitalet, Denmark
Other Study IDs: H-24051777; p-2024-17691 (Other: Privacy, Capital Region of Denmark)
Record Dates: First submitted 2026-01-06; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Acute Brain Injury; Hydrocephalus; External Ventricular Drain; External Ventricular Drainage Associated Infection
MeSH Terms: conditions — Brain Injuries; Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sampling of blood and cerebrospinal fluid — As soon as possible after placement of the external drain, and then in intervals of 1-3 days;
  * CSF analyses: cerebrospinal fluid group analysis (eosinophilic granulocytes, erythrocytes, glucose, nucleated cells, leucocytes (mononuclear), lymphocytes, macrophages, monocytes, neutrophil granulocytes, protein, and smudge cells) and lactate (L-lactate and D-lactate). Analyses will be performed by the Dept. of Biochemistry, Rigshospitalet, Denmark.
  * CSF microscopy and culture: Analysed by the Dept. of Microbiology, Rigshospitalet, Denmark.
  * Blood: C-reactive protein, differentials (leukocytes, neutrophile granulocytes, erythrocytes, lymphocytes). Analyses will be performed by the Dept. of Biochemistry, Rigshospitalet, Denmark.
  * Blood: lactate and glucose. Point of care (POC) analysis by blood gas analyser (Radiometer ABL800 Series Flex Q, Denmark)

SUMMARY:
This observational study involving patients with acute brain injury undergoing treatment with an external ventricular drain consists of three subprojects, aiming to:

1. investigate various biomarkers, with a primary focus on the development of cerebrospinal fluid lactate in relation to ventriculostomy-associated infection;
2. compare proximal and distal sample results obtained from an external ventricular drain;
3. describe the natural progression of various biomarkers in blood and cerebrospinal fluid following acute brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* EVD in situ
* Admission to the neuro-ICU or neurosurgical step-down unit at Rigshospitalet, Denmark
* Diagnosis of acute brain injury categorized as traumatic brain injury, subarachnoid haemorrhage, intracranial haemorrage, intraventricular haemorrhage

Exclusion Criteria:

* Patient or closest relatives do not understand written and spoken Danish or English
* Patients transferred to Rigshospitalet with an EVD
* Patients with brain injury due to existing brain infection (e.g., meningitis, intracranial empyema or abscess, encephalitis)
* Patients with existing ventriculoperitoneal or ventriculoatrial shunt at the time of admission
* Patients with primary or secondary brain cancer
* Patients died or in palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute brain injury, that are treated with an external ventricular drain
Sampling Method: Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of cerebrospinal fluid lactate | Throughout the external ventricular drain duration (1-60 days)
  in patients with compared to patients without positive CSF culture, and for b. patients with both a positive CSF culture and a distinct drop in the level of consciousness compared to patients with negative CSF culture and a stable level of consciousness.

SECONDARY OUTCOMES:
CSF lactate concentration change in patients developing ventriculostomy associated infection | Throughout the external ventricular drain duration (1-60 days)
  Concentration of CSF lactate and other CSF markers a. before, during and after detection of organisms in patients with a positive CSF culture, and b. if no organisms are detected, during the first, second and third tertile of EVD treatment.
Functional outcome at six months | 6 months after the initial brain injury
  Functional outcome evaluated six months after the initial brain injury using:
  1) modified Rankin Scale (mRS) as favourable (0-2) or unfavourable (3-6)
Functional outcome at six months | 6 months after the initial brain injury
  Functional outcome evaluated six months after the initial brain injury using:
  2) Glascow Outcome Score-Extended (GOS-E) as favorable (5-8) or unfavorable (0-4)
Comparison of concentration of cerebrospinal fluid markers drawn from the proximal and distal port of the EVD | Throughout the external ventricular drain duration (1-60 days)
  Mean difference, limits of agreement, intraclass correlation, mean of absolute difference and consistency between measurements of CSF markers drawn from the proximal and distal port of the EVD.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
IPD will only be shared with a data sharing agreement